CLINICAL TRIAL: NCT05897957
Title: Continued Evaluation of Patients With Parkinson's Disease Who Previously Received BRT-DA01, a Human Embryonic Stem Cell-Derived Midbrain Dopaminergic Neuronal Cell Therapy
Brief Title: Continued Evaluation of Patients With Parkinson's Disease Who Previously Received BRT-DA01
Status: Enrolling by invitation | Type: Observational
Sponsor: BlueRock Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BRT-DA01-501
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biomarkers for PD may be explored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter study to evaluate the safety and clinical outcomes of BRT-DA01 in subjects with PD who previously received BRT-DA01 in the Phase 1 Study MSK-DA01-101.No investigational therapy will be administered in this study.

DETAILED DESCRIPTION:
All subjects who received BRT-DA01 transplantation in Study MSK-DA01-101 (ie, parent study) will be asked to enroll in Study BRT-DA01-501. Subjects enrolled in this study are to be monitored for safety and clinical outcomes through 5 years post-BRT-DA01 transplantation. For individual participating subjects, the Baseline visit for the BRT-DA01-501 study will be defined as the last observation recorded in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Subject received BRT-DA01 in Study MSK-DA01-101 (ie, parent study) and will have completed or discontinued the parent study
* Subject must be willing and able to provide written informed consent for the BRT-DA0-501 study in accordance with applicable regulations and guidelines and to comply with all study visits and procedures

Exclusion Criteria:

* No exclusion criteria

Ages: 50 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson's Disease who previously received BRT-DA01 in the Phase 1 Study MSK-DA01-101
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total SAEs and total number of subjects with at least 1 SAE | Baseline through 5 years post-transplantation
  Total SAEs and total number of subjects with at least 1 SAE related to cellular drug product

SECONDARY OUTCOMES:
Change in striatal 18F-DOPA uptake using positron emission tomography (PET) | Baseline through 5 years post-transplantation
  Change in striatal 18F-DOPA uptake using positron emission tomography (PET)
Change in Hauser PD diary measurements | Baseline through 5 years post-transplantation
  Change in Hauser PD diary measurements
Change in the International Parkinson and Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline through 5 years post-transplantation
  Change in the MDS-UPDRS
Change in levodopa equivalent daily dose (LEDD) | Baseline through 5 years post-transplantation
  Change in LEDD
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) summary index | Baseline through 5 years post-transplantation
  Change in PDQ-39
Change in the Unified Dyskinesia Rating Scale (UDysRS) | Baseline through 5 years post-transplantation
  Change in UDysRS

OTHER OUTCOMES:
Adverse Events | Baseline through 5 years post-transplantation
  AEs related to the cellular drug product
Change in modified Schwab and England Activities of Daily Living (mSEADL) scale | Baseline through 5 years post-transplantation
  Change in mSEADL
Change in brain atrophy using MRI | Baseline through 5 years post-transplantation
  Change in brain atrophy using MRI
Subjects using alternative advanced treatment options in Parkin's Disease | Baseline through 5 years post-transplantation
  Number of subjects using alternative advanced treatment options in PD (eg, CSAI, LCIG, DBS, focused ultrasound ablation)

CONTACTS AND LOCATIONS:
Overall Officials: Nauman Abid, MD, Study Director — BlueRock Therapeutics LP
Locations (3):
- United States (2):
  - University of California, Irvine, Orange, California
  - Weill Cornell Medical College, New York, New York
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No